CLINICAL TRIAL: NCT01890499
Title: PROSPECTIVE RANDOMIZED CONTROLLED TRIAL ON CLEAR FEEDS VERSUS LOW RESIDUE DIET AFTER SURGERY IN ELECTIVE COLORECTAL SURGERY PATIENTS.
Brief Title: Prospective Controlled Trial On Clear Feeds Versus Low Residue Diet After Surgery In Elective Colorectal Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Fleshner MD, Program Director, Colorectal Surgery Fellowship Shierley, Jesslyne, and Emmeline Widjaja Chair in Colorectal Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00029966
Record Dates: First submitted 2013-06-27; First posted 2013-07-01 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Nausea/Vomiting
Keywords: tolerability; diet after operation
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low residue diet arm (Experimental): Two arm randomized controlled trial. First arm is the Clear feeds on postoperative day one arm.
  The second arm (interventional arm) is the Low Residue diet on postoperative day one arm.
  Interventions: Dietary Supplement: Low Residue diet arm.
- Clear feeds arm (Active Comparator): Standard of care is to start clear feeds on postoperative day one for elective colorectal surgery patients.
  Interventions: Dietary Supplement: Low Residue diet arm.

INTERVENTIONS:
Dietary Supplement: Low Residue diet arm. — Interventional arm is to provide low residue diet on postoperative day one.

SUMMARY:
Prospective randomized controlled trial investigating commencement of low residue diet versus clear feeds on postoperative day one following elective colorectal surgery, with regards to patient tolerability, incidence of nausea and/or vomiting, and postoperative length of hospitalization stay.

DETAILED DESCRIPTION:
Based on current literature, the incidence of postoperative nausea and vomiting varies widely and can reach up to 40% in abdominal surgery patients. Thus, patient tolerability to postoperative enteral feeds is taken as 60%. This is a superiority trial: group one is the clear feeds group and patient tolerability in this group is taken to be 60%. Group two is the low residue diet group.

The primary hypothesis is that the incidence of postoperative ileus is not affected by the consistency of enteral diet given, and patients who are placed on low residue diet from postoperative day one do not have an increased risk of postoperative nausea and vomiting as compared to patients who are placed on clear feeds.

The primary endpoint measured is Patient tolerability, as evidenced by development of vomiting on postoperative day two.

Key Inclusion criteria are:

1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
2. Males or females, >18 years of age inclusive at the time of study screening;
3. American Society of Anesthesiologists (ASA) Class I-III;
4. Colorectal surgery (open and/or laparoscopic);
5. Elective Surgery.

Key Exclusion criteria are:

1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures.
2. Children <18 years of age.
3. Pre-operative clinical diagnosis of intestinal obstruction.
4. Pre-existing known upper gastrointestinal disorders.
5. Pre-existing oropharyngeal disorders such as stomatitis, altered taste sensations.
6. Open upper abdominal surgical incisions.
7. Colorectal surgery with concomitant resectional surgery of the stomach or proximal jejunum (small bowel).
8. Pregnant patients.
9. Bedbound or moribund patients.
10. Pre-existing history of clinical depression.
11. Epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
2. Males or females, >18 years of age inclusive at the time of study screening;
3. American Society of Anesthesiologists (ASA) Class I-III;
4. Colorectal surgery (open and/or laparoscopic);
5. Elective Surgery.

Exclusion Criteria:

1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures.
2. Children <18 years of age.
3. Pre-operative clinical diagnosis of intestinal obstruction.
4. Pre-existing known upper gastrointestinal disorders.
5. Pre-existing oropharyngeal disorders such as stomatitis, altered taste sensations.
6. Open upper abdominal surgical incisions.
7. Colorectal surgery with concomitant resectional surgery of the stomach or proximal jejunum (small bowel).
8. Pregnant patients.
9. Bedbound or moribund patients.
10. Pre-existing history of clinical depression.
11. Epidural analgesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Development of nausea and vomiting on postoperative day two | postoperative day two

CONTACTS AND LOCATIONS:
Overall Officials: philip R Fleshner, M.D, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States